CLINICAL TRIAL: NCT03967236
Title: Impact of Intestinal Virome on Pediatric Inflammatory Bowel Disease
Acronym: IVOIRE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0794
Record Dates: First submitted 2019-05-23; First posted 2019-05-30 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and blood samples from paediatric inflammatory bowel disease patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of stool and blood samples — For each visit, stool and blood samples will be collected during a pediatric gastroenterology day hospital stay.
  This collection of stool and blood specific IVOIRE study is carried out in the context of examination already planned for the usual care of the patient.

SUMMARY:
Over the last few years, dysbiosis has emerged as a possible trigger of gut inflammation in inflammatory bowel disease (IBD) and a promising therapeutic target. The complex diversity of microbiota was initially highlighted by the powerful new tools in genetics, including next-generation sequencing (NGS). NGS permitted to decipher the composition of bacterial intestinal communities, but also that of the gut virome. Since then, the evidence of a dynamic instability of the enteric virome in IBD has grown considerably. IBD patients present an expansion of bacteriophages (Caudovirales) associated with decreased bacterial diversity. Moreover, gut virome richness seems to differ between Crohn's disease (CD) and ulcerative colitis (UC) patients. These insights open the gate of new diagnostic, predictive, and therapeutic approaches. However, little is known about pediatric IBD gut virome in terms of variability and evolution under the influence of different treatments (exclusive enteral nutrition, immunosuppressive therapy and biologics). The aim of this study is to evaluate the gut family viral diversity and relative abundance of eukaryotes and prokaryotes in paediatric IBD patients

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-17 years
* Follow-up in pediatric gastroenterology for inflammatory bowel disease :

  * Crohn's disease
  * Hemorrhagic rectocolitis
* Introduction of anti-TNFa treatment in the Pediatric Gastroenterology Day Hospital of the "Hôpital Femme Mère Enfant" service in Lyon
* Collection of the non-opposition of at least one of the holders of the parental authority present and the child in the medical file

Exclusion Criteria:

* Refusal to participate in the study
* Antibiotherapy in the 4 weeks preceding the sampling
* Patient with ileostomy or colostomy.
* Patient who has undergone extensive bowel resection.
* History of intestinal surgery (except appendectomy)
* Patient subject to a legal protection measure

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with nflammatory bowel disease newly treated with anti-TNF therapy in the "Hôpital Femme Mère Enfant" center in Lyon
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluation over time of change of the gut virome | at the inclusion, 6 months and one year
  Abundance measure: number of sequences generated for a given family or species.
  Viral isolation, extraction, and amplification of viral nucleic acids from patient's stools.
  Next generation sequencing Statistical analysis
Evaluation over time of change of the gut virome | at the inclusion, 6 months and one year
  Measure of relative abundance: abundance of a given family or species relative to other species or families in the sample.
  eukaryote versus prokaryote virus
  Viral isolation, extraction, and amplification of viral nucleic acids from patient's stools.
  Next generation sequencing Statistical analysis
Evaluation over time of change of the gut virome | at the inclusion, 6 months and one year
  Measure of alpha diversity by the Shannon index which takes into account the number of species present, but also the distribution of these species.
  Viral isolation, extraction, and amplification of viral nucleic acids from patient's stools.
  Next generation sequencing Statistical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Service de gastroentérologie nutrition, hépatologie pédiatrique - Hôpital Femme Mère Enfant groupement hospitalier Est - HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No